CLINICAL TRIAL: NCT01735032
Title: Contribution of Multimodal Imaging (MRI, PET, MEG) in Pre-surgical Evaluation of Drug-resistant Focal Epilepsy
Brief Title: Multimodal Imaging in Pre-surgical Evaluation of Epilepsy
Acronym: EPIMAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-703
Record Dates: First submitted 2012-10-22; First posted 2012-11-28 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-10

CONDITIONS: Partial Epilepsy
Keywords: focal epilepsy; pre-surgical evaluation; multimodal imaging; SEEG
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Epilepsy is the most common chronic neurological disorder in the world, affecting more than 50 million people worldwide. Approximately 35% of patients with epilepsy are refractory to all available antiepileptic drugs. Drug-resistant epilepsies are often partial or focal. Patients with drug-resistant focal epilepsy suffer from an increased risk of death, primarily due to seizure-related fatalities, in comparison with the general population. The only therapeutic option for this form of epilepsy is the surgical removal of the region of the brain responsible for seizures, called the epileptogenic zone (EZ). This requires the precise localization of the EZ based on a comprehensive pre-surgical evaluation of patients.

Today the gold standard for localizing the EZ and validating a non-invasive technique for localization of the EZ remains intracerebral stereo-EEG (stereo-electroencephalography or SEEG) recordings of spontaneous seizures. The implementation strategy of the intracerebral depth electrodes is guided by clinical and neuroimaging data, including anatomical Magnetic Resonance Imaging (MRI), Positron Emission Tomography (PET) with FDG (fluoro-Deoxy-Glucose) and MagnetoEncephaloGraphy (MEG). Although the contribution of each technique in the pre-surgical localization of the EZ has already been shown, no wide-scale study has examined the cumulative contribution of these three techniques.

DETAILED DESCRIPTION:
The purpose of this study is (i) to evaluate rigorously the diagnostic value of multimodal imaging for non-invasive localization of the EZ and (ii) to better target the indications for intracerebral recordings (SEEG).

ELIGIBILITY:
Inclusion Criteria:

* Patient with drug-resistant focal epilepsy
* Candidates for pre-surgical evaluation including FDG PET, MRI, MEG and SEEG recordings.
* Age 18-65 years
* EEG-confirmed focal epilepsy for >2 years
* Signed informed consent form.

Exclusion Criteria:

* Age <18 years and >65 years
* Contraindication to the MRI
* Pregnant woman
* Head size incompatible with MEG recordings
* Adult subject to legal protection measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with drug-resistant focal epilepsy and candidates for epilepsy surgery will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-11 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Localizing value of MEG, FDG-PET and MRI for the determination of the Epileptogenic Zone defined by SEEG recordings | 180 days
  Pathological volumes defined by multimodal imaging (MEG, FDG-PET and MRI) will be compared to the topography of the EZ defined by SEEG recordings.
  For each patient, we will sum the total number of intracerebral depth electrodes included in the EZ. Then, for each functional volume obtained from multimodal data fusion, we will count the total number of electrodes in the latter (Vol elec_tot) and the number of electrodes included in the EZ (Vol elec_ze).

SECONDARY OUTCOMES:
sensitivity and specificity | 180 days
  For each functional volume, two parameters will be defined: sensitivity and specificity. These parameters will be calculated as follows: sensitivity = (Vol elec_ze) / (Pat elec_ze) and specificity = (Vol elec_ze) / (Vol elec_tot).

CONTACTS AND LOCATIONS:
Overall Officials: François MAUGUIERE, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France